CLINICAL TRIAL: NCT01150409
Title: Hemodynamic and Inflammatory Effects of Abrupt Versus Tapered Corticosteroid Discontinuation in Septic Shock
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting eligible subjects
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-336
Record Dates: First submitted 2010-06-21; First posted 2010-06-25 (Estimated); Results first posted 2015-09-02 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Septic Shock
Keywords: Sepsis; hydrocortisone
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Hydrocortisone; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydrocortisone (Experimental): Hydrocortisone 50 mg IV every 12 hours x 4 doses (2 days), followed by Hydrocortisone 50 mg IV every 24 hours x 2 doses (2 days)
  Interventions: Drug: hydrocortisone; Drug: Normal Saline
- Normal Saline (placebo) (Placebo Comparator): 0.9% sodium chloride (equal volume to hydrocortisone) IV every 12 hours x 4 doses (2-days), followed by 0.9% sodium chloride (equal volume to hydrocortisone) IV every 24 hours x 2 doses (2-days)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: hydrocortisone — 1) Hydrocortisone 50 mg IV every 12 hours x 4 doses (2 days), followed by Hydrocortisone 50 mg IV every 24 hours x 2 doses (2 days)
  Other Names: 11β,17α,21-trihydroxypregn-4-ene-3,20-dione
  Arms: hydrocortisone
Drug: Normal Saline — 0.9% sodium chloride (equal volume to hydrocortisone) IV every 12 hours x 4 doses (2-days), followed by 0.9% sodium chloride (equal volume to hydrocortisone) IV every 24 hours x 2 doses (2-days)
  Other Names: 0.9% sodium chloride

SUMMARY:
The proposed study will evaluate the potential benefit of a tapered course of hydrocortisone compared to abrupt cessation in patients initiated on hydrocortisone for septic shock. The study will include adult patients in the medical intensive care unit (MICU) who meet criteria for corticosteroid therapy for septic shock according to the current MICU protocol.All patients will receive 7 days of hydrocortisone (50mg/Q6hrs) as part of the routine management of septic shock, before being randomly assigned to receive hydrocortisone taper versus no taper. The primary study endpoint is the incidence of hypotension within 7 days after randomization. Secondary endpoints will include incidence of adrenal insufficiency, and changes in the inflammatory status (assessed by cytokine measurements) before, during, and after corticosteroid discontinuation. The cytokines to be measured include IL-1, IL-6, IL-9, IL-10, and TNF. Since there has not been a randomized clinical trial to investigate the potential benefit of weaning septic patients off low-dose hydrocortisone as opposed to stopping abruptly, this study has potential to change clinical practice by leading to a consistent approach of corticosteroid discontinuation and to a better understanding of their impact on the inflammatory modulation in septic shock.

DETAILED DESCRIPTION:
Current therapy for septic shock includes antimicrobials, fluid resuscitation, catecholamines, and measures to improve tissue oxygen delivery. The use of corticosteroids as an adjunctive treatment in septic shock has been an area of intensive research over the past decade. A handful of studies suggest that patients in septic shock benefit from low-dose glucocorticoids.Low-dose corticosteroids may improve hemodynamics, decrease vasopressor requirements, and reduce 28-day mortality in patients with vasopressor-refractory septic shock. A meta-analysis from 2004 also suggested that the use of low-dose corticosteroids does not significantly increase the risk of superimposed infections, gastrointestinal bleeding, or hyperglycemia.

The exact mechanism for this beneficial effect has not been completely established, although direct vascular effects and anti-inflammatory effects of corticosteroids have been proposed. While there is ongoing debate over which subpopulations of patients derive benefit from corticosteroids, there is as much controversy regarding the appropriate duration of therapy. The current Surviving Sepsis Campaign suggests that intravenous IV hydrocortisone 200-300mg/day should be given to adult septic shock patients after it has been confirmed that their blood pressure is poorly responsive to fluid resuscitation and vasopressor therapy. The duration of therapy is not specified. There is also no clear evidence to suggest that patients benefit from tapering steroids as opposed to stopping them abruptly; both strategies have been employed. Annane showed both a mortality benefit and shorter duration of vasopressor therapy with an abrupt end to a 7-day course of hydrocortisone and fludrocortisone in patients with septic shock compared to placebo; while others showed a similar benefit with a taper.Keh demonstrated reversal of both hemodynamic and immunologic effects after a three-day treatment of "low-dose" hydrocortisone, suggesting that some of the beneficial effects of steroids disappear in less than 24 hours. Interestingly, 30% of patients had to restart vasopressor therapy after discontinuation of corticosteroids in one of the Keh's study arms.

ELIGIBILITY:
Inclusion Criteria:Patients who meet the following criteria will be enrolled in the study:

* suspected septic shock
* initiation of hydrocortisone 50mg IV Q6H (per MICU protocol)
* written informed consent signed by patient or legal surrogate
* Septic shock is defined by meeting all of the following requirements:
* Clinical evidence of infection. Clinical evidence of infection is defined as the presence of a known or probable source of infection that has necessitated the initiation of systemic antimicrobial therapy. Clinical evidence of infection could include (but is not limited to) one or more of the following:

  1. presence of increased number of PMNs (neutrophils) in normally sterile body fluid
  2. positive culture or gram stain of blood, sputum, urine, or normally sterile body for a pathogenic microorganism
  3. chest radiograph consistent with a diagnosis of pneumonia with a positive culture, gram stain, diagnostic bronchoalveolar lavage, or protected specimen brush for a respiratory tract pathogen
  4. focus of infection identified by visual inspection (e.g., ruptured bowel found at surgery, wound with purulent drainage, radiographic or Computed tomographic evidence of an abscess or osteomyelitis, etc.) and
  5. patient has an underlying disease or condition that is highly likely to be associated with infection (e.g., ascending cholangitis, ischemic bowel, etc.)
* Two of the following:

  1. Core temperature either > 38°C (> 100.4°F) or < 36°C (< 96.8°F)
  2. Tachycardia. Heart rate greater > 90 beats/minute
  3. Respiratory rate > 20 b/min or PaCO2 < 32 torr, or need for mechanical ventilation due to sepsis
  4. WBC > 12 or < 4 K/mm3
* End-organ cardiovascular dysfunction defined as hypotension unresponsive to fluid replacement necessitating vasopressor therapy, or lactate ≥4 mmol/L

Exclusion Criteria:

* age less than 18
* previous systemic corticosteroid therapy in the past 90 days (prednisone >5 mg/d or equivalent)
* pregnancy
* Acquired Immune Deficiency Syndrome (AIDS)
* hematological malignancies
* advanced form of cancer with less than 30-day life expectancy
* patients who receive fludrocortisone
* evidence of prior acute myocardial infarction

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Guzman, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocortisone | Normal Saline (Placebo)
Started | 11 | 0
Completed | 11 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult MICU pateints who meet criteria for corticosteroid therapy of septic shock
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone | Normal Saline (Placebo) | Total
Number analyzed (Participants) | 11 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 9 |  | 9
  >=65 years | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 |  | 5
  Male | 6 |  | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hypotension Between Study Days 8 and 14 (Within 7 Days of the Initiation of Study Drug).
Description: Study screening/enrollment stopped due to lack of eligible subjects. No outcome measures were analyzed due to the low enrollment.
Time Frame: Day 14
Arm/Group | Hydrocortisone | Normal Saline (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Hydrocortisone | Normal Saline (Placebo)
Serious Adverse Events (participants affected / at risk) | 9/11 | 0/0
Other Adverse Events (participants affected / at risk) | 0/11 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone (N=11) | Normal Saline (Placebo) (N=0)
Septic Shock/Multi System Organ Failure (General disorders) | 2 (2) | 0 (0)
Septic Shock/Poor Prognosis/Family Reuest to Withdraw Support (General disorders) | 2 (2) | 0 (0)
End Stage Liver Disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Respiratory Failure (General disorders) | 1 (1) | 0 (0)
ARDS/H1N1 (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes